CLINICAL TRIAL: NCT03063879
Title: Efficacy and Safety of Sofosbuvir and Daclatasvir in Treating Patients With Hepatitis C and Renal Failure.
Brief Title: Treating Hepatitis C in CRF Using Sofosbuvir and Daclatasvir
Acronym: SD-CRF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Ahvaz Jundishapur University of Medical Sciences (Other); Shiraz University of Medical Sciences (Other); Hamadan University of Medical Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 96-04-37-37348
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2018-02

CONDITIONS: Hepatitis C, Chronic; Chronic Renal Failure
Keywords: hepatitis C; renal failure; sofosbuvir; daclatasvir
MeSH Terms: conditions — Hepatitis C, Chronic; Kidney Failure, Chronic; Hepatitis C; Renal Insufficiency | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sovodak (Experimental): Sofosbuvir 400 mg and daclatasvir 60 mg
  Interventions: Drug: Sofosbuvir 400 mg and daclatasvir 60 mg

INTERVENTIONS:
Drug: Sofosbuvir 400 mg and daclatasvir 60 mg — Daily fixed dose combination pill (Sovodak) containing 400 mg sofosbuvir and 60 mg daclatasvir for 12 weeks if not cirrhotic (liver stiffness < 12 KPa) or 24 weeks if cirrhotic
  Other Names: Sovodak

SUMMARY:
Sofosbuvir is the base of most treatment regimens for hepatitis C. In patients with renal failure the blood level of one of its metabolites (GS-331007) rises up to 20 folds. Although no particular adverse event has been linked to this metabolite sofosbuvir is not recommended for patients with renal failure mainly because of lack of data. Nevertheless there are anecdotal reports and small studies proving the safety of sofosbuvir in renal failure. This study addresses this lack of information by evaluating the safety and efficacy of sofosbuvir and daclatasvir in treating hepatitis C in 100 patients with renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Positive qualitative hepatitis C virus RNA test on two occasions at least 6 months apart
* Renal failure (eGFR < 30 cc/min) or under hemodialysis

Exclusion Criteria:

* Model for End-stage Liver Disease (MELD) score > 20,
* Child's C (CTP score > 12),
* Heart rate < 50/min,
* Taking amiodarone

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sustained Viral Response (SVR12) | 12 weeks after end of treatment
  Lack of detectable hepatitis C virus in blood 12 weeks after end of treatment

SECONDARY OUTCOMES:
Safety as assessed by adverse drug events | From start of treatment to 12 weeks after end of treatment
  Adverse drug events recorded by direct questioning

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Merat, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Shariati Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poustchi H, Majd Jabbari S, Merat S, Sharifi AH, Shayesteh AA, Shayesteh E, Minakari M, Fattahi MR, Moini M, Roozbeh F, Mansour-Ghanaei F, Afshar B, Mokhtare M, Amiriani T, Sofian M, Somi MH, Agah S, Maleki I, Latifnia M, Fattahi Abdizadeh M, Hormati A, Khoshnia M, Sohrabi M, Malekzadeh Z, Merat D, Malekzadeh R. The combination of sofosbuvir and daclatasvir is effective and safe in treating patients with hepatitis C and severe renal impairment. J Gastroenterol Hepatol. 2020 Sep;35(9):1590-1594. doi: 10.1111/jgh.14994. Epub 2020 Feb 5. PMID 31994788